CLINICAL TRIAL: NCT02965209
Title: European Novel Motorized Spiral Endoscopy Trial
Acronym: ENMSET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Evangelisches Krankenhaus Düsseldorf (Other)
Collaborators: Olympus (Industry)
Responsible Party: Principal Investigator, Torsten Beyna, MD, Evangelisches Krankenhaus Düsseldorf
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENMSET
Record Dates: First submitted 2016-11-11; First posted 2016-11-16 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Disorder of Small Intestine; Gastrointestinal Hemorrhage; Iron Deficiency Anaemia; Crohn's Disease; Small Bowel Tumors; Intestinal Polyposis Syndrome; Coeliac Disease
Keywords: endoscopy; small bowel endoscopy; motorized spiral endoscopy; spiral endoscopy
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Anemia, Iron-Deficiency; Crohn Disease; Celiac Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- motorized spiral enteroscopy (Experimental): Novel Motorized Spiral Enteroscopy (NMSE) represents a new technology which offers all of the advantageous options of spiral enteroscopy with a faster and less invasive approach.
  Interventions: Procedure: motorized spiral enteroscopy

INTERVENTIONS:
Procedure: motorized spiral enteroscopy — Novel Motorized Spiral Enteroscopy (NMSE) represents a new technology which offers all of the advantageous options of spiral enteroscopy with a faster and less invasive approach. When the region of interest in the small bowel is reached by NMSE standard endoscopic techniques, e.g. argon plasma coagulation (APC), forceps biopsy or endoscopic mucosal resection (EMR) are performed for treatment and/or tissue acquisition.
  Other Names: standard endoscopic interventions (not experimental)

SUMMARY:
The subject Novel Motorized Spiral Enteroscope (NMSE) represents a new technology which offers all of the advantageous options of spiral enteroscopy with a faster and less invasive approach. The system is similar to other currently marketed endoscopes in that it incorporates a flexible insertion tube, light source, digital imaging, and channels for passing accessories for sample collection or therapeutic interventions. The NMSE system is unique in that it incorporates a user-controlled motor contained in the endoscope's handle to rotate a spiral cuff located on the endoscope's insertion tube. Rotation of this cuff, which has soft spiral-shaped "fins", pleats the small bowel on to the endoscope's insertion tube, thereby allowing rapid and atraumatic access deep into the small bowel. The system also includes a display monitor, a motor control unit, device to display measured motor current and signal torque, and a set of foot pedals. Motorization of the Spiral Enteroscope and limitation of rotation to a short cuff instead of a long overtube promise to accelerate the procedure, to facilitate insertion and to improve maneuvering the instrument in comparison to conventional spiral enteroscopy

DETAILED DESCRIPTION:
General anesthesia and/or sedation will be prescribed according to institutional practices and clinical judgment; type, amount and duration will be recorded.

A standard esophagogastroduodenoscopy (EGD) will be performed prior to the enteroscopy. If during this preliminary exam the endoscopist identifies any stricture or believes the patient has anatomy that would cause excessive resistance during Novel Motorized Spiral insertion or examination, the patient will be withdrawn from the study and the reason for study withdrawal will be noted.

The Novel Motorized Spiral endoscope will be inserted and advanced with the assistance of motorized clockwise spiral rotation, (controlled directly by the operating physician via the foot pedal). If at any point a stricture is observed or excessive resistance to the advancement of the endoscope is encountered, further advancement of the endoscope must cease and the reason for procedure termination documented on the case report form.

After reaching the depth of insertion required for patient treatment or diagnosis, the endoscope will be withdrawn using motorized counter-clockwise spiral rotation, also controlled by the foot pedal. Maximum depth of insertion will be recorded as the maximum insertion depth when failure to advance the endoscope tip after repositioning the patient, applying abdominal pressure and/or using other standard measures fails to advance the endoscope OR the investigator decides to terminate advancement based on clinical judgment. During withdrawal, the endoscopist will cumulatively estimate the length of bowel released from the endoscope tip in order to calculate the total depth of insertion. Insertion depth will be referenced to the Ligament Treitz. If the clinician decides to mark the point of maximum insertion, the tissue may be tattooed by first creating a saline bleb, followed by the injection of India ink (e.g., SPOT).

Tissue sampling and/or therapies will be performed during withdrawal as clinically appropriate. The details of all sampling and/or therapies (number, type & location) will be recorded.

The comfort and cardiopulmonary stability of the patient will be monitored throughout the procedure, as per the standard of care - this includes continuous pulse oximetry, blood pressure, and heart rate monitoring.

Photographs or video recordings are used to document any significant lesions and any tissue trauma.

Postprocedural measures Patients will be hospitalized for at least 24 hours after NMSE because of the potential risk of delayed adverse events. Only liquid diet is allowed during the first 12 hours in asymptomatic patients. Clinical investigation and determination of the blood cell count and the serum level of C-reactive protein will be done after 24 hours. 30 days after the procedure patients will be interviewed by a telephone call for evaluation of complaints or delayed complications. Discomfort (location and severity (0-10 VAS) should be documented immediately after NMSE, after 24 hours and before discharge.

ELIGIBILITY:
Inclusion Criteria:

* Overt obscure gastrointestinal bleeding or obscure gastrointestinal bleeding or indeterminate iron-deficiency anaemia and positive videocapsule endoscopy (VCE) or negative VCE in patients who have ongoing bleeding shown by overt bleeding or continued need for blood transfusions
* Abdominal pain or chronic diarrhoea with positive findings of small bowel imaging examinations
* Noncontributory ileocolonoscopy and suspicion of Crohn's disease on small-bowel cross-sectional imaging modalities or small-bowel capsule endoscopy
* Further evaluation of known Crohn's disease or therapeutic indications in Crohn's disease
* Imaging tests suspicious for small-bowel tumour
* Large polyps (>10-15mm) discovered by radiological examination or small-bowel capsule endoscopy in patients with Peutz-Jeghers syndrome
* Nonresponsive or refractory coeliac disease

Exclusion Criteria:

* Age under 18 years
* Health status American Society of Anesthesiologists classification (ASA) 4
* Pregnancy
* Coagulopathy (INR≥2.0, Platelets < 70/nl)
* Taking anti-platelet agents or anticoagulants (other than aspirin) within last 7 days
* Any medical contraindication to standard enteroscopy
* Presence of any intraluminal or extraluminal foreign body in the abdominal cavity
* Any prior gastric, small bowel or colonic surgery, or implantable devices in these locations (cardiac pacemakers and non-abdominal implants are acceptable)
* Known or suspected bowel obstruction or stenosis or history of bowel obstruction
* Known coagulation disorder
* Known or suspected esophageal stricture or Schatzki ring
* Known gastric or esophageal varices
* Suspected perforation of the GI tract
* Inability to tolerate sedation or general anesthesia for any reason
* Inability to tolerate endotracheal intubation
* Absence of a signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2015-11; Primary Completion 2018-02-03 (Actual); Study Completion 2018-02-06 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield of NMSE in patients with suspected small bowel diseases | 30 days

SECONDARY OUTCOMES:
Procedural success | 30 days
Procedural time (minutes) | 30 days
Depth of maximal insertion (cm) | 30 days
Therapeutic yield | 30 days
Adverse events | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Horst Neuhaus, MD, Principal Investigator — Evangelisches Krankenhaus Duesseldorf
Locations (2):
- Universite Libre des Bruxelles, Brussels, Belgium
- Evangelisches Krankenhaus, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Beyna T, Arvanitakis M, Schneider M, Gerges C, Boing D, Deviere J, Neuhaus H. Motorised spiral enteroscopy: first prospective clinical feasibility study. Gut. 2021 Feb;70(2):261-267. doi: 10.1136/gutjnl-2019-319908. Epub 2020 Apr 24. PMID 32332141